CLINICAL TRIAL: NCT01029587
Title: Eculizumab to Enable Renal Transplantation in Patients With History of Antiphospholipid Antibody Syndrome or Catastrophic Antiphospholipid Antibody Syndrome
Brief Title: Eculizumab to Enable Renal Transplantation in Patients With History of Catastrophic Antiphospholipid Antibody Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NA_00029904
Record Dates: First submitted 2009-12-09; First posted 2009-12-10 (Estimated); Results first posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Antiphospholipid Antibody Syndrome; End Stage Renal Disease
Keywords: CAPS; Kidney transplant; Renal transplant; Catastrophic Antiphospholipid Antibody Syndrome
MeSH Terms: conditions — Antiphospholipid Syndrome; Kidney Failure, Chronic | interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eculizumab (Experimental): Patients will receive eculizumab in conjunction with systemic anticoagulation before and after kidney transplant operation
  Interventions: Drug: Eculizumab

INTERVENTIONS:
Drug: Eculizumab — Eculizumab will be administered by intravenous infusion. Eculizumab will be administered at a dose of 1200mg by intravenous (IV) infusion on the day of or on the day prior to kidney transplantation, and at a dose of 900mg IV on post-operative day 1. Subsequently, the post-operative dosing regimen would be comprised of an induction phase of weekly doses of 900mg IV per dose followed by a maintenance phase of every other week dosing of 1200mg IV per dose. The weekly induction dosing regimen would begin on postoperative day 8, and would continue for three doses (specifically, doses of 900mg IV would be given on postoperative days 8, 15, and 22). The maintenance phase of dosing would begin with a dose of 1200mg on postoperative day 29, and would continue for a total of 5 doses (specifically, doses of 1200mg IV would be given on postoperative days 29, 43, 47, 72, and 85). In most cases, eculizumab would be discontinued after the 5th maintenance dose.
  Other Names: Soliris

SUMMARY:
Catastrophic Antiphospholipid Antibody Syndrome (CAPS) is a rare condition in which life-threatening blood clots form in multiple organs simultaneously and can lead to multi-organ system failure and death. The causes of CAPS are not entirely understood, but CAPS episodes are often triggered by stressful events such as infections, surgery, or trauma. For patients who survive an episode of CAPS, permanent kidney failure is not uncommon because the kidneys are the organ system most frequently affected in CAPS. Kidney transplantation is the treatment of choice for end-stage kidney disease, but patients with a history of CAPS are exceptionally high-risk kidney transplant recipients because the chance that surgery itself could trigger a life-threatening or transplant-threatening episode of CAPS is significant. As a result, patients with CAPS are not generally considered candidates for transplantation. Despite this, these patients have a severely decreased life-expectancy on dialysis and their long-term survival and quality of life would be greatly increased by a successful kidney transplant. In this trial, a drug called eculizumab will be tested for its ability to prevent CAPS after kidney transplantation in patients with a prior history of CAPS. Eculizumab is an inhibitor of the complement system, which is believed to be important in generating the inflammatory environment that leads to diffuse clotting of blood vessels in CAPS. The investigators hypothesize that by blocking the complement cascade using eculizumab, in conjunction with blocking the coagulation system, that kidney transplantation can be safely and successfully performed in patients with a history of CAPS.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* History of Catastrophic Antiphospholipid Antibody Syndrome (CAPS)
* End-stage renal disease

Exclusion Criteria:

* Any contraindications to transplantation other than CAPS
* Pregnant women
* Women who intend to become pregnant over the study period
* Ongoing or untreated meningococcal infections
* History of serious adverse reaction to eculizumab

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2010-05-06 (Actual); Study Completion 2010-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Philosophe, MD, PHD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Eculizumab
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Eculizumab
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Prevention of Catastrophic Antiphospholipid Antibody Syndrome (CAPS) After Kidney Transplant
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 1
Participants | 1

2. Secondary Outcome: Number of Patients With Kidney Transplant Graft Survival
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 1
Participants | 1

3. Secondary Outcome: Number of Patients Who Survive
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Eculizumab
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eculizumab (N=1)
neutropenia (Immune system disorders) | 1 (1)
subtherapeutic INR (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No